CLINICAL TRIAL: NCT01567995
Title: Randomised, Double-blind, Placebo-controlled Study of Topical Clobetasone Butyrate Cream in Patients With Eczema for Two Weeks to Evaluate the Efficacy and Safety
Brief Title: Randomised, Double-blind, Placebo-controlled Study of Topical Clobetasone Butyrate 0.05% Cream in Subjects With Eczema for Two Weeks to Evaluate the Efficacy and Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111187
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Eczema
Keywords: eczematous; dermatitis
MeSH Terms: conditions — Eczema; Dermatitis | interventions — clobetasone butyrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clobetasone Butyrate 0.05% Cream (Experimental): Clobetasone Butyrate 0.05% Cream
  Interventions: Drug: Clobetasone Butyrate 0.05% Cream
- Vehicle (base cream) (Other): Vehicle (base cream)
  Interventions: Drug: Vehicle (base cream)

INTERVENTIONS:
Drug: Clobetasone Butyrate 0.05% Cream — Clobetasone Butyrate 0.05% Cream
  Arms: Clobetasone Butyrate 0.05% Cream
Drug: Vehicle (base cream) — Vehicle (base cream)
  Arms: Vehicle (base cream)

SUMMARY:
This was a multicenter, randomised, double-blind, two treatment arms, vehicle (cream base) -controlled, parallel-group study in subjects with moderate to severe eczema (defined by investigators global assessment (IGA) score greater than or equal to 3).

Subjects were screened within 3 days prior to randomization. At the screen visit, subjects gave informed consent and were then assessed for health status and eligibility for inclusion in the study. At the baseline visit, subject eligibility was assessed for randomization (Day 0). Eligible subjects were randomised to Clobetasone Butyrate 0.05% Cream group or vehicle (cream base) group at the rate of 1:1. During the treatment phase, subjects returned to the sites in day 7 post-baseline visit for assessment of their disease status and eligibility to continue on the study. During the final visit, 14 days after the baseline, subjects returned to the study sites for assessment of their disease status before completing the study. In addition, the safety and tolerability of Clobetasone Butyrate 0.05% cream were also assessed through the whole trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of eczema, fulfil the 3 follow items: 1) Erythema, papilla/water blister, Lichenification, skin damage with infiltration, 2) unknown reason, recurrent attacks; 3) itching in diseased skin
* Subjects must have body surface area (BSA) disease involvement of less than or equal to 10% as assessed by palm method
* Subject must present with moderate and above eczema as defined by a score greater than or equal to 3 using the investigators global assessment (IGA) of eczema severity.

Exclusion Criteria:

* The subject presents with any systemic disorder or active skin disease (e.g. psoriasis) that would in any way confound interpretation of the study results or subjects who present with scars, moles, tattoos, body piercings, sunburn in the test area which could interfere with the assessment of lesions at screening.
* The subject has eczema restricted to the face, the feet or the hands only.
* The subject is indicated any anti-infectives drug for a current complication of overt bacterial, fungal and viral infection
* History of recent (<1 month) active or presence of current superficial skin infections of viral aetiology such as herpes simplex, or varicella.
* The subject has been exposed to below therapy within the set timeframe: Topical agents administered in the diseased skin, including emollient - 1 week; Systemic administration of anti-histamine agents - 2 week; Systemic administration of corticosteroid -4 week; Systemic administration of immunosuppressive drugs - 4 week; UV therapy -4 week
* Foreseeable intensive ultraviolet (UV) exposure during the study (solar or artificial). Subjects must not be exposed to intense direct sunlight for long periods, and must not use skin tanning devices (e.g. sunbed) for the duration of the study.
* History of clinically significant cardiovascular, pulmonary, gastrointestinal, liver, neurological, renal or haematological abnormalities.
* History of allergy to components of test medications to be used in the study.
* History of anaphylaxis (a sudden, potentially life-threatening systemic allergic reaction) to food, medications, insect venom, or latex.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-02-28 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2009-02-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Eczema Area and Severity Index (EASI) score at Day 7 | Baseline, Day 7
  Investigators assessed presence and severity of erythema, induration/papulation, excoriation, and lichenification in four body areas using EASI: head/neck, upper limbs, trunk, and lower limbs. Investigators assigned a severity score from 0 - 3 for each area (none=0, mild=1, moderate=2, and severe=3). Investigators also assigned an area score from 0 (no eruption) to 6 (>90-100% eruption) for each area. The weighting factor was 0.1 for head/neck, 0.2 for upper limbs, 0.3 for trunk, and 0.4 for lower limbs. The total body score for each body region was obtained by multiplying the sum of the severity scores of the four key signs by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gave the EASI total, ranging from 0 to 72. A higher score represented greater disease severity. A negative change from baseline indicates improvement.
Change from baseline in Eczema Area and Severity Index (EASI) score at Day 14 | Baseline, Day 14
  Investigators assessed presence and severity of erythema, induration/papulation, excoriation, and lichenification in four body areas using EASI: head/neck, upper limbs, trunk, and lower limbs. Investigators assigned a severity score from 0 - 3 for each area (none=0, mild=1, moderate=2, and severe=3). Investigators also assigned an area score from 0 (no eruption) to 6 (>90-100% eruption) for each area. The weighting factor was 0.1 for head/neck, 0.2 for upper limbs, 0.3 for trunk, and 0.4 for lower limbs. The total body score for each body region was obtained by multiplying the sum of the severity scores of the four key signs by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gave the EASI total, ranging from 0 to 72. A higher score represented greater disease severity. A negative change from baseline indicates improvement.
Reduction Percentage of Eczema Area and Severity Index (EASI) score after 7 day of treatment | up to Day 7
  Investigator assessed surface & severity of erythema, induration/papulation, excoriation & lichenification in four body areas using EASI: head/neck, upper extremities, trunk & lower extremities. Investigators assigned a severity score (0-3) for each area (none=0, mild=1, moderate=2, severe=3). Investigators also assigned an area score from 0 (no eruption) to 6 (>90-100% eruption) for each area. Weighting factor was 0.1 for head/neck, 0.2 for upper extremities, 0.3 for trunk & 0.4 for lower extremities. Total body score for each body region was obtained by multiplying sum of severity scores by area score, then multiplying result by constant weighted value assigned to that body region. Sum of these scores gave EASI total, ranging from 0 to 72. Reduction percentage of score was calculated as: (sum of score after day 7 minus sum of score at baseline) *100/sum of score after day 7. Lesser negative reduction percentage lesser severity of disease, more effectiveness of treatment.
Reduction Percentage of Eczema Area and Severity Index (EASI) score after 14 days of treatment | up to Day 14
  Investigator assessed surface & severity of erythema, induration/papulation, excoriation & lichenification in four body areas using EASI: head/neck, upper extremities, trunk & lower extremities. Investigators assigned a severity score (0-3) for each area (none=0, mild=1, moderate=2, severe=3). Investigators also assigned an area score from 0 (no eruption) to 6 (>90-100% eruption) for each area. Weighting factor was 0.1 for head/neck, 0.2 for upper extremities, 0.3 for trunk & 0.4 for lower extremities. Total body score for each body region was obtained by multiplying sum of severity scores by area score, then multiplying result by constant weighted value assigned to that body region. Sum of these scores gave EASI total, ranging from 0 to 72. Reduction percentage of score was calculated as: (sum of score after day 14 minus sum of score at baseline) *100/sum of score after day 14. Lesser negative reduction percentage lesser severity of disease, more effectiveness of treatment.

SECONDARY OUTCOMES:
Change from baseline in Investigators Global Assessment (IGA) graded score at Day 7 and Day 14 | Baseline, Day 7 and Day 14
  The IGA was used to determine disease severity in a given time and describe severity of eczema using scale of 0 to 6 as follows: 0 Clear:=No inflammatory signs of eczema; 1 Almost clear=Just perceptible erythema and just perceptible papulation/infiltration; 2 Mild:=Mild erythema and mild papulation/infiltration; 3 Moderate:=Moderate erythema, and moderate papulation/infiltration; 4 Severe= Severe erythema, and severe papulation/infiltration; 5 Very Severe=Very severe erythema, and very severe papulation/infiltration with oozing/crusting. Lesser score indicate lesser disease severity.
Changes from baseline in Visual Analog Scale (VAS) at Day 7 and Day 14 | Baseline, Day 7 and Day 14
  Participants assessed the degree of their pruritus using a 100-mm visual analog scale (VAS; 0mm=No itch, 100mm=maximum itch) at Baseline, Day 7 and Day 14. Higher pruritus/itch VAS score indicating more severe pruritus/itching.
Number of participants with participants-based assessment score of disease control at Day 7 and Day 14 | Day 7 and Day 14
  The participant's assessment score is a semi-quantitative score intended to reflect the participants own evaluation of disease control. It consisted of a four-point scale ranging from complete disease control (0) to uncontrolled disease (3): 0 - Complete disease control; 1 - Good disease control; 2 - Limited disease control; 3 - Uncontrolled disease. Lesser score indicate better disease control.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- China (4):
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin